CLINICAL TRIAL: NCT04584476
Title: Superior Capsular Reconstruction Versus. Partial Repair for Irreparable Rotator Cuff Tears: A Prospective Comparative Study
Brief Title: Superior Capsular Reconstruction Versus. Partial Repair for Irreparable Rotator Cuff Tears
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Chunyan Jiang, Director of Sports Medicine Service of Beijing Jishuitan hospital, Beijing Jishuitan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CJiang-SCR
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Rotator Cuff Tears
Keywords: Irreparable Rotator Cuff Tears; Superior Capsular Reconstruction
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCR group (Experimental): underwent superior capsular reconstruction
  Interventions: Procedure: superior capsular reconstuction
- Partial group (Other): underwent partial rotator cuff repair
  Interventions: Procedure: partial rotator cuff repair

INTERVENTIONS:
Procedure: superior capsular reconstuction — these patients underwent arthroscopic superior capsular reconstuction
  Arms: SCR group
Procedure: partial rotator cuff repair — these patients underwent arthroscopic partial rotator cuff repair
  Arms: Partial group

SUMMARY:
Rotator cuff tear is one of the common injuries that cause shoulder pain in the elderly. After the rotator cuff tendon is injured, repairing the torn rotator cuff tendon through arthroscopic surgery is an effective treatment that is currently widely used. In the rotator cuff injury, irreparable rotator cuff injury is a difficult point in treatment, especially for patients with a long injury time, the obvious shrinkage of the injured tendon, muscle atrophy and steatosis may occur, all of which lead to the poor quality of the rotator cuff tendon needed to be repaired , Poor healing ability, seriously affecting the shoulder joint function and daily life of these patients. For this part of patients, arthroscopic partial repair of torn rotator cuffs is one of the commonly used methods. In addition, in recent years, superior capsular reconstruction has been gradually applied to the clinic and has achieved good clinical effects, but there are no controlled studies to compare Clinical effect of partial repair and superior capsular reconstruction on irreparable rotator cuff injury.

ELIGIBILITY:
Inclusion Criteria:

* patients with Irreparable Rotator Cuff Tears
* underwent superior capsular reconstruction or partial repair
* at least two years follow-up

Exclusion Criteria:

* reparable Rotator Cuff Tears
* underwent reverse total shoulder arthroplasty

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons (ASES) score | 2 year postoperatively
  A patient-reported outcome measurement
Acromiohumeral distance (AHD) | 1 year postoperatively
  measured in x-ray
retear rate | 1 year postoperatively
  measured in MRI

CONTACTS AND LOCATIONS:
Overall Officials: Chunyan Jiang, Principal Investigator — Sports Medicine Service, Beijing Jishuitan hospital

IPD SHARING:
Plan to Share IPD: No